CLINICAL TRIAL: NCT03261752
Title: Investigating the Role of SPG20,STK31 Genes in the Carcinogenesis of Colorectal Cancer
Brief Title: New Genes in the Carcinogenesis of Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariana Anwar, Demonstrator of cancer biology, Assiut University
Other Study IDs: CRC
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient with cancer: blood sample will be collected from patient before and after treatment (surgery or chemotherapy)
  Interventions: Diagnostic Test: blood sample
- healthy people: blood sample will be collected for comparison
  Interventions: Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: blood sample — Total genomic DNA will be extracted DNA extraction kit using a QIAamp DNA Blood Mini kit .Genetic analysis of both SPG20 &STK31 by RTPCR.

SUMMARY:
Colo rectal cancer is one of the greatest ,mutual malignancies worldwide ,accounting for an estimated 1.3 million new cases and >500,000 mortality ⁄ year . is the fourth leading cause of cancer-associated mortality worldwide with speedily ,cumulative ,occurrence rate in the worldwide

DETAILED DESCRIPTION:
colo rectal cancer represents a global and local problem, as it is one of the commonest types of cancer all over the world. Globally, Colo rectal cancer in women (9.2% of diagnoses) it is the second most common cause of cancer . it is the third most common in men (10.0%). After lung, stomach, and liver cancer it is the fourth most common cause of cancer death.

Cancer is a multistep procedure resulting from an ongoing accretion of genetic and epigenetic fluctuations to the genome.

Spartin is a protein that in humans is encoded by the SPG20 gene. This protein may be involved in endosomal trafficking, microtubule dynamics, or both functions. Aberrant promoter methylation of genes is a common epigenetic alteration in colo rectal cancer .

This has stimulated the prospect to implement a dependable, reasonable and simple approach for Colo rectal detection . The SPG20 gene is situated in chromosome band 13q13.3; the SPG20 gene converts the spartin protein, which is a multi functional protein that has formerly been recognized to be complicated in intra cellular epidermal growth factor receptor trading , The serine-threonine kinase 31 (STK31) gene was initially identified through cDNA subtraction as a testis-specific protein kinase gene expressed in mouse spermatogonia . Recently, STK31 has been described as a novel cancer testis (CT) antigen, highly expressed in Gastrointestinal cancer cells (colo rectal, gastric and esophageal cancer), while restricted to testis and fetal brain in normal tissues .

It was found that SPG20 is mutated in Troy er syndrome, an hereditary spastic paraplegia

ELIGIBILITY:
Inclusion Criteria:

* age between 35-65
* patient with colorectal cancer (at any stage)
* both sex included

Exclusion Criteria:

* pediatric patients
* patient with insufficient data
* cardiac patient
* pregnant women

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient between 35-65 who are newly diagnosed with colorectal cancer
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
detection of SPG20&STK31 genes | 5 months
  detection of SPG20&STK31 genes and prediction future treatment for colo-rectal cancer